CLINICAL TRIAL: NCT01539564
Title: Multi-Center Phase 3 Trial of Minocycline HCl 1mg Microspheres for the Use in Subjects With Peri-Implantitis
Brief Title: Arestin - Use in Subjects With Peri-Implantitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OraPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-P-5267
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Treatment (minocycline HCl microspheres, 1mg) administered at Baseline (following randomization) and Day 90 to qualifying implant sites, plus full-mouth mechanical debridement (deep cleaning) at Baseline and Day 180.
  Interventions: Drug: Minocycline HCl Microspheres
- Control (No Intervention): Full-mouth mechanical debridement (deep cleaning) at Baseline and Day 180; no treatment

INTERVENTIONS:
Drug: Minocycline HCl Microspheres
  Other Names: Arestin (brand name)
  Arms: Treatment

SUMMARY:
The objective of the study is to evaluate the safety and effectiveness of Arestin (minocycline HCl) 1 mg Microspheres in the treatment of subjects with peri-implantitis, when used in combination with mechanical debridement.

The hypothesis of the study is that Arestin in combination with mechanical debridement is more effective in the treatment of peri-implantitis when compared to mechanical debridement alone. The primary efficacy measure will be the reduction of probing depth at Day 180 as measured at qualifying implant sites.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of one osseointegrated implant with a diagnosis of peri-implantitis
* Absence of any significant oral soft tissue pathology
* At least one peri-implant site with an average of 2 probing depth readings between 5mm and 7mm (inclusive) when using a light force and with bleeding on probing within 30 seconds of the probing
* Confirmed evidence of pathologic bone loss
* At least 1mm of keratinized gingiva present around the implant

Exclusion Criteria:

* Pregnancy
* Allergy to tetracycline-class drug(s)
* Systemic medical condition(s) requiring antibiotic prophylaxis prior to invasive dental procedures
* Presence of active systemic infectious disease such as hepatitis, HIV, history of tuberculosis
* Diagnosis of clinically significant or unstable organic disease, or compromised healing potential
* Signs of untreated advanced periodontal disease and/or poor oral hygiene
* Subjects having a probing depth greater than 8mm at time of enrollment
* Subjects presenting with mobility of any dental implant
* Subjects having a qualifying implant under occlusal trauma or overloaded (as determined by the investigator)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in mean Probing Depth of qualifying implant sites | Baseline to Day 180

SECONDARY OUTCOMES:
Change in percentage of qualifying implants with Bleeding on Probing | Baseline to Day 180
Change in mean Probing Depth of qualifying implant sites | Baseline to Day 90
Change in percentage of qualifying implants with Bleeding on Probing | Baseline to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Flemmig, DMD, MBA, Principal Investigator — University of Washington, School of Dentistry
Locations (12):
- United States (9):
  - UCLA School of Dentistry - Oral and Maxillofacial Surgery, Los Angeles, California
  - University of Florida College of Dentistry, Gainsville, Florida
  - Georgia Regents University, Augusta, Georgia
  - University of Maryland, School of Dentistry, Baltimore, Maryland
  - University of Minnesota - School of Dentistry, Minneapolis, Minnesota
  - University of North Carolina, General Oral Health Center, Chapel Hill, North Carolina
  - Ohio State University College of Dentistry, Columbus, Ohio
  - The Periodontal-Implant Institute, McLean, Virginia
  - University of Washington, School of Dentistry, Seattle, Washington
- University of Dusseldorf, Poliklinik fur Zahnerhaltung, Parodontologie und Endodontologie, Düsseldorf, Germany
- Kristianstad University, Department of Periodontology, Kristianstad, Sweden
- Eastman Dental Institute, University College of London, London, United Kingdom